CLINICAL TRIAL: NCT05287373
Title: Clinical Study Of a Micro-Implantable Pulse Generator For The Treatment of Peripheral Neuropathic Pain
Acronym: COMFORT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nalu Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NAL-01-2021-US
Record Dates: First submitted 2022-02-08; First posted 2022-03-18 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Neuralgia; Chronic Pain
Keywords: PNS; Peripheral nerve stimulation; mIPG; peripheral nerve stimulator
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PNS Therapy plus Conventional Medical Management (Active Comparator): peripheral nerve stimulator plus conventional medical management
  Interventions: Device: Nalu Neurostimulation System for PNS; Other: conventional medical management
- Conventional Medical Management (Other): Control arm conventional medical management only
  Interventions: Other: conventional medical management

INTERVENTIONS:
Device: Nalu Neurostimulation System for PNS — The Nalu Neurostimulation System for PNS is a peripheral nerve stimulator
  Other Names: Nalu PNS
  Arms: PNS Therapy plus Conventional Medical Management
Other: conventional medical management — Conventional medical management

SUMMARY:
This post market study is being conducted to document the comparative effectiveness and safety of peripheral nerve stimulation plus conventional medical management versus conventional medical management alone in the treatment of chronic, intractable peripheral neuralgia of post-traumatic or post-surgical origin. This is a prospective, minimal risk, multi-center, randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18 to 80 years of age at the time of enrollment.
2. Subject would have been prescribed PNS therapy regardless of participation in this study; the use of the Nalu device must be on-label.
3. Subject has been diagnosed with one or more of the conditions listed below in the low back, shoulder, knee, or foot (including ankle):Post-surgical/post-traumatic peripheral neuralgia including but not limited to pain due to peripheral nerve injury, post-surgical scar formation, nerve entrapment; Mononeuropathy, specified or unspecified or in diseases classified elsewhere; Other neuralgia or neuropathic pain; Osteoarthritic pain.
4. Subject has chronic (defined as at least 6 months duration), intractable peripheral neuropathic pain, exclusive of the craniofacial region; any nociceptive pain must be less prominent than the neuropathic pain. Pain should have a predominant neuropathic component as per the investigator's clinical assessment.
5. Subject should have a pain score of at least 6, in the target area of pain, as recorded on the BPI-Q5 (NRS) at screening.
6. Subject is willing to cooperate with the study requirements including, compliance with the study procedures and completion of all study visits.
7. Subject reported stable pain (non-escalating) for 60 days prior to signing informed consent.
8. Subject is currently receiving CMM and has had stable pain medication use and dosage for 30 days prior to signing informed consent.
9. Subject is psychologically qualified to receive a peripheral nerve stimulator as per the clinician's standard clinical practice and judgment and does not have clinically relevant psychological condition(s) that would interfere with their ability to accurately report outcomes or complete study procedures.
10. Subject has demonstrated the ability to appropriately place the adhesive clip in the location where the IPG is most likely to be implanted. Alternatively, subject is able to appropriately use the relief belt and/or limb cuff to keep the Therapy Disc in place.

Exclusion Criteria:

1. Subject currently has an active implantable medical device such as a drug pump, spinal cord stimulator, peripheral nerve stimulator, sacral nerve stimulator, deep brain stimulator, and/or cardiac pacemaker.
2. Subject has previously failed PNS or Spinal Cord Stimulation (SCS) or Dorsal Root Ganglion (DRG) therapy (trial or permanent implant)
3. Pain is completely absent at rest.
4. Patient has clinical evidence of complex regional pain syndrome (CRPS), peripheral neuralgia of metabolic origin, post-herpetic neuralgia, biochemical evidence of a metabolic or genetic neuropathy (e.g., Charcot'- Marie- Tooth Disease) or mixed motor/sensory polyneuropathy.
5. Subject has a medical condition that would prevent them from participating in the current study per investigator's or medical monitor's judgment.
6. Subject has had a successful (≥ 50% pain relief) interventional procedure within the past 3 months to treat the same pain condition(s) being examined in this study including, nerve blocks.
7. Uncontrolled depression or uncontrolled psychiatric disorders
8. Subject is currently participating in another clinical investigation with an active treatment arm.
9. Subject is allergic or sensitive to materials used in the device components including, skin adhesives or does not tolerate the wearable aspect of the device.
10. Subject has pending or ongoing legal issues (including unresolved worker's compensation claims or equivalent) or other conflicting secondary gain issues related to their chronic pain condition.
11. Subject has a current diagnosis of a coagulation disorder, bleeding diathesis, or progressive peripheral vascular disease that has not been medically corrected.
12. Subject has an active systemic infection.
13. Subject is unable to read and/or write in English or give informed consent.
14. Subject has a life expectancy of less than 1 year.
15. Subject has an active malignant neoplasm (metastatic or local) or evidence of paraneoplastic syndrome.
16. Subject with uncontrolled diabetes mellitus, showing signs of diabetic neuropathy, as evidenced by a neurological exam and a HbA1c test.
17. Subject has evidence of an alcohol or drug dependency within the last 6 months prior to enrollment.
18. Subject is pregnant (if female and sexually active, subject must be using a reliable form of birth control, be surgically sterile or be at least 1 year post-menopausal).
19. Subject is nursing/breastfeeding.
20. Subject is on ≥90 mg-morphine equivalents per 24 hours.
21. Subject has undergone an ablative treatment of the target peripheral nerve, or proximal nerve trunk giving rise to the target nerve, or dorsal roots (and DRGs) that ultimately make up the target nerve. No ablative procedures directed at the spinal cord, dorsal roots, or peripheral nerve(s) being treated in the study. To note, subjects who have undergone RF ablation of the dorsal rami, cool pulsed RF of the facet innervation may be considered for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness: Responder rates between groups | 3-months
  Difference in responder rates between groups. Responder rate is defined as the percent of subjects with 50% or greater pain relief from baseline, based on the BPI-Q5 (NRS).
Safety: Rate of serious and non-serious adverse events between groups | 3-months
  Rate of serious and non-serious adverse events between groups

SECONDARY OUTCOMES:
Responder Rates between groups at 6-months | 6 months
  Difference in responder rates between groups. Responder rate is defined as the percent of subjects with 50% or greater pain relief from baseline, based on the BPI-Q5 (NRS).
Responder Rates between groups at 12-months | 12-months
  Difference in responder rates between groups. Responder rate is defined as the percent of subjects with 50% or greater pain relief from baseline, based on the BPI-Q5 (NRS).
Responder Rates between groups at 24-months | 24-months
  Difference in responder rates between groups. Responder rate is defined as the percent of subjects with 50% or greater pain relief from baseline, based on the BPI-Q5 (NRS).
Responder Rates between groups at 36-months | 36-months
  Difference in responder rates between groups. Responder rate is defined as the percent of subjects with 50% or greater pain relief from baseline, based on the BPI-Q5 (NRS).
Functional Outcomes: Change in ODI, BDI, EQ-5D, BPI from baseline | 3, 6, 9, 12, 18, 24, 30 and 36 months
  Change in patient reported outcomes from baseline between groups
Safety Assessment | 3, 6, 9, 12, 18, 24, 30 and 36 months
  Rate of serious and non-serious events

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Martin, Study Director — Nalu Medical
Locations (5):
- United States (5):
  - Arizona Pain Specialists, Scottsdale, Arizona
  - Denver Back Pain Specialists, Greenwood Village, Colorado
  - International Spine, Pain and Performance Center, Washington D.C., District of Columbia
  - Institute of Precision Pain Medicine, Corpus Christi, Texas
  - Northwest Pain Care, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hatheway J, Hersel A, Engle M, Gutierrez G, Khemlani V, Kapural L, Moore G, Ajakwe R, Trainor D, Hah J, Staats PS, Makous J, Heit G, Kottalgi S, Desai MJ; COMFORT Study Group. Clinical study of a micro-implantable pulse generator for the treatment of peripheral neuropathic pain: 12-month results from the COMFORT-randomized controlled trial. Reg Anesth Pain Med. 2024 Nov 20:rapm-2024-106099. doi: 10.1136/rapm-2024-106099. Online ahead of print. PMID 39572166